CLINICAL TRIAL: NCT04947358
Title: Longitudinal Observational Study for mIddle Term Follow-up Patients Admitted for Acute Dyspnea in TunIsia
Acronym: SIDI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: S Form Pharma (Industry)
Responsible Party: Sponsor
Other Study IDs: AD201801
Record Dates: First submitted 2019-07-19; First posted 2021-07-01 (Actual); Last update posted 2021-07-01 (Actual); Status verified 2021-06

CONDITIONS: Longitudinal Observational Study With 6 Months Follow-up

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of the SIDI study is to follow, few months after discharge from the hospital, the patients admitted to the 3 emergency departments in Tunisia for acute dyspnea and to determine the proportion and the factors favoring rehospitalization and death.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted for unexpected respiratory difficulty
* Patient admitted to the emergency department
* One of the following 3 criteria have to be present at admission to the ER:
* O2 < or = 95%
* Respiratory rate RR > or = 20
* Suffocation sensation

Exclusion Criteria:

* Patients <18 years old and> 85 years' old
* Pregnancy
* History of allergic asthma at early age
* Diagnosis retained of pulmonary embolism
* Patients with heart failure (HF) with left ventricular ejection fraction LVEF <40% are known beforehand or discovered at admission to ER
* known Allergy for Polyamide; Polyester; Elastane; Silicone; Silver; Synthetic material Cardiorespiratory disorders which may be aggravated by the slight compression of the thorax Open wound on the skin, at the level of the trunk

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients admitted for unexpected respiratory difficulty
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2019-02-22 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Proportion and causes of re-hospitalization and deaths within 3 months of discharge from hospital | 3 months
  Define the proportion and causes of re-hospitalization and deaths within 3 months of discharge from hospital for patients admitted to the Emergency Department for acute dyspnea

SECONDARY OUTCOMES:
Proportion and causes of re-hospitalization and deaths within 6 months of discharge from hospital | 6 months
  Check theses parameters at 6 months, differentiating the cardiac causes from non-cardiac causes and the effect of home follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- ER, Fattouma Bourguiba Hospital, Monastir, Tunisia

IPD SHARING:
Plan to Share IPD: Undecided